CLINICAL TRIAL: NCT01727531
Title: IDO2 Genetic Status Informs the Neoadjuvant Efficacy of Chloroquine in Brain Metastasis Radiotherapy.
Brief Title: IDO2 Genetic Status Informs the Neoadjuvant Efficacy of Chloroquine (CQ) in Brain Metastasis Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Health (Other)
Responsible Party: Principal Investigator, Albert DeNittis, Principal Investigator, Main Line Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R09-2775L
Record Dates: First submitted 2012-11-07; First posted 2012-11-16 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Brain Metastasis
Keywords: chloroquine; WBRT; survival; brain metastasis; radiotherapy; SNPs; gene coding; immunoregulatory enzyme IDO2
MeSH Terms: conditions — Brain Neoplasms | interventions — chloroquine diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CQ Arm (Experimental): 250 mg chloroquine once a day by mouth beginning one week prior to beginning radiation therapy and continue for a total of five weeks.
  Interventions: Drug: Chloroquine diphosphate

INTERVENTIONS:
Drug: Chloroquine diphosphate — 250 mg chloroquine once a day by mouth beginning one week prior to beginning radiation therapy and continue for a total of five weeks

SUMMARY:
This research is being done to determine if a short course of Chloroquine (five weeks) before, during and after whole brain radiation therapy (WBRT) will improve the overall survival of subjects being treated for brain metastases.

DETAILED DESCRIPTION:
Hypothesis one: A short course of chloroquine one week prior and four weeks after initiation of WBRT is tolerable and significantly increases the median survival time of patients suffering from brain metastasis as assessed one, three, six, nine, twelve and 24 months post radiotherapy, when compared to historic controls.

Hypothesis two: The presence of one or both single-nucleotide polymorphisms (SNP)s in the gene coding for the immunoregulatory enzyme indoleamine 2,3-dioxygenase 2 (IDO2) improves the clinical outcomes of WBRT or the response to CQ co-treatment.

3.2. Specific Aims:

The specific aims of this study are:

1. Determine patients physical profiles prior WBRT and at regular intervals afterwards up to 24 months after radiotherapy.
2. Record the status of patient metastases (i.e. number, location, size)
3. Determine patients' KPS values.
4. Record the incidence and causes of mortality of patients.
5. Determine the genotype of IDO2 for each patient.
6. Following data analysis, test the validity of the two hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed primary solid malignancy
* Patients with single or multiple brain metastases
* Patients with metastasis diameter < 5 cm
* Age > 18
* Clearance from the patient's physician that treatment with chloroquine should not pose a problem to the patient

Exclusion Criteria:

* Patients with a history of hypotension, cardiomyopathy, epilepsy, seizures
* Patients with impaired renal function
* Patients with psoriasis, porphyria
* Patients with known hypersensitivity to 4-aminoquinoline compounds
* Pregnancy, nursing
* Prior radiotherapy
* During the chloroquine treatment, patients complaining from visual or auditory disturbances, and patients suffering from acute gastrointestinal problems i.e. Anorexia, nausea, vomiting, diarrhea, abdominal cramps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Specific Aim | up to 24-months after completion of treatment
  Determine patients physical profiles prior WBRT and at regular intervals afterwards up to 24 months after radiotherapy

SECONDARY OUTCOMES:
Secondary endpoint: death | up to 24 months after completion of treatment
  from any cause

OTHER OUTCOMES:
Additional Aims | up to 24 months after completion of treatment
  Record the status of patient metastases (i.e. number, location, size)
Additional Aims | up to 24 months after completion of treatment
  Record KPS
Additional Aims | up to 24 months after completion of treatment
  Record genotype of IDO2

CONTACTS AND LOCATIONS:
Overall Officials: Albert DeNittis, MD, Principal Investigator — Main Line Health
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States